CLINICAL TRIAL: NCT03900507
Title: Postoperative Results of Patients Who Received Medical Treatment for Incisional Endometriosis and Did Not Respond to Treatment
Brief Title: Postoperative Results of Incisional Endometriosis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, M.D, Department of Obstetrics and GynecologyR, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.11.44
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Endometriosis; Pain
Keywords: incisional endometriosis; scar endometriosis
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endometriosis surgery — Medical treatment was initiated in patients with abdominal incision due to endometriotic focus in the incision line.
  however, patients with surgical excision indications were the study group.

SUMMARY:
The primary aim is to determine the endometriotic foci formed in the incision line after surgical operations, and the medical treatment approach is the primary objective. Medical treatment was initiated and the patients who did not benefit from the treatment would be operated and postoperative pain scores would be compared with the medical treatment. It will be tried to determine which treatment is more effective in pain control.

In addition to removing the symptoms and providing therapeutic methods in patients, it is aimed to help in differential diagnosis of dermatological diseases and malignancy and thus to prevent anxiety in patients. It is also aimed to evaluate the pathology results in the most appropriate way to eliminate the symptoms (severe pain, bleeding, etc.) that occur in accordance with the menstrual cycle every month.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone surgery previously and who have an incision in the abdominal region and who applied with a complaint of mass in the incision and who were primarily considered endometrial focus in the diagnosis,
* Patients who were diagnosed with endometriotic foci in the incision line and used medical treatment for a while, but who did not benefit because of surgical excision.

Exclusion Criteria:

* Dermatologically diagnosed patients
* Follow-up patients with malignancy diagnosis
* Patients who have responded to medical treatment

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patients who have undergone surgery previously and who have an incision in the abdominal region and who applied with a complaint of mass in the incision and who were primarily considered endometrial focus in the diagnosis,
  -Patients who were diagnosed with endometriotic foci in the incision line and used medical treatment for a while, but who did not benefit because of surgical excision.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
preoperative pain scores | 1 week
  The preoperative pain scores of the patients who were planned for operation due to incisional endometriosis and who were more likely to receive medical treatment will be evaluated with visuel visual scale (vas).
  vas score '0' no pain; The vas score '10' will be recorded as unbearable pain.
postoperative pain scores | 1 week
  The postoperative pain scores of the patients who were planned for operation due to incisional endometriosis and who were more likely to receive medical treatment will be evaluated with visuel visual scale (vas).
  vas score '0' no pain; The vas score '10' will be recorded as unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)